CLINICAL TRIAL: NCT00588224
Title: Validation and Application of 3-dimensional Ultrasound for Measurement of Gastric Volumes in Healthy Subjects
Brief Title: 3D Ultrasound Validation for Measuring Stomach Volume
Acronym: 3DUSstomach
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Michael Camilleri MD, Mayo Clinic
Other Study IDs: 07-005231
Record Dates: First submitted 2007-12-22; First posted 2008-01-08 (Estimated); Last update posted 2009-07-22 (Estimated); Status verified 2009-07

CONDITIONS: Healthy
Keywords: stomach; accommodation; volume; SPECT; 3 dimensional ultrasonography; healthy volunteers

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: adults
  Interventions: Other: 3D ultrasound
- 2: adolescents
  Interventions: Other: 3D ultrasound

INTERVENTIONS:
Other: 3D ultrasound — measurement of stomach volume by 3D ultrasound

SUMMARY:
The goal is to study the accuracy of 3-dimensional ultrasound (which does not involve radiation) to measure the size of the stomach, comparing it with a previously validated method that involves radiation. This will make it possible to check the stomach function of children without exposing them to radiation. A second goal is to measure the size of the stomach and the effect of a standard meal on stomach volume in adolescent boys and girls.

DETAILED DESCRIPTION:
Specific Aims

1. To compare the fasting and postprandial volumes measured by 99mTc- SPECT (standard test) and 3-D ultrasound in 12 healthy adults in order to test latter's external validity
2. To assess the performance characteristics of 3-D ultrasound for the measurement of gastric volumes during fasting and in response to a standard meal, specifically, the intra- and inter-individual coefficient of variation in 12 healthy adults who undergo two estimations of fasting and postprandial volumes
3. To develop normative data for fasting and postprandial gastric volumes in 24 asymptomatic adolescents.

Study Design

The study will be conducted in 2 parts: first, 12 healthy adults will undergo SPECT and 3-D ultrasound in random order (aim 1); one week after the first ultrasound examination, a second Ultrasound examination will be conducted in all participants (aim 2) In the second part, 24 adolescents (12 in each gender, 12 aged 13-15, 12 aged 16-18)) will undergo a single determination of fasting and postprandial gastric volumes during fasting and post-prandially. The methods and validation of the SPECT study have been previously published (2). Three D ultrasonography will be conducted using state of the art equipment following methods published in the literature. (3)

The study will screen 80 healthy adults or adolescents in order to enroll 12 healthy adulkts for the first two aims, and 24 adolescent healthy subjects for the third aim.

For subjects in group 1, the order of SPECT and 3D- ultrasound tests will be randomized.

The randomization assignments will be made according to a pre-study schedule prepared by the Section of Biostatistics. Medical investigators will be blinded to assignment, allocation will be concealed

ELIGIBILITY:
Inclusion Criteria:

1. Age: 13-65 years
2. Body mass index (BMI): 18 to 32 (exept in adolescents)
3. Negative urine pregnancy test for women of childbearing potential
4. Absence of gastrointestinal symptoms (abridged Bowel Disease Questionnaire)
5. Signed informed consent

Exclusion Criteria:

1. Subjects with body mass index (BMI) of less than 18 or more than 32.
2. Structural or metabolic diseases/conditions that affect the gastrointestinal system, or functional gastrointestinal disorders. For screening, the Bowel Disease Questionnaire will be used to exclude subjects with irritable bowel syndrome.
3. Use of drugs or agents within the past 2 weeks that alter GI transit including laxatives, magnesium or aluminum-containing antacids, prokinetics, erythromycin, narcotics, anticholinergics, tricyclic antidepressants, SSRI and newer antidepressants.

   NOTE: Low stable doses of thyroid replacement, estrogen replacement, low dose aspirin for cardioprotection, and birth control pills or depot injections are permissible.
4. Female subjects who are pregnant or breast feeding.
5. Females must be either surgically sterilized, postmenopausal (>12 months since last menses) or, if of childbearing potential, using reliable methods of contraception as determined by the physician (single-barrier methods alone and rhythm methods are not acceptable).
6. Clinical evidence (including physical exam and ECG) of significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematological, neurological, psychiatric, or other disease that interfere with the objectives of the study. Any candidate participants with such disorder mentioned will be referred to their general physician.
7. Symptoms of a significant clinical illness in the preceding two weeks.
8. Participation in another clinical study within the past 30 days.
9. Subjects who are considered by the investigator to be alcoholics not in remission or known substance abusers.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: ealthy adolescents and adults: The study will screen up to 80 healthy adults or adolescents in order to enroll 12 healthy adults for the first two aims, and 24 adolescent healthy subjects for the third aim
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2007-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Fasting and Postprandial gastric volumes measured by 3D ultrasonography in adults and adolescents | one month

SECONDARY OUTCOMES:
Intra and inter-individual COV in adults for fasting and postprandial volumes | one month
Accuracy of 3D-ultrasonography in measurement of fasting and posprandial volume using Bland-Altman plot | one month

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Camilleri, MD, Principal Investigator — Mayo Clinic